CLINICAL TRIAL: NCT03944512
Title: A Randomized Controlled Trial of Pravastatin to Prevent Preeclampsia in High Risk Women
Brief Title: Pravastatin to Prevent Preeclampsia
Acronym: Pravastatin
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: participants are no longer being examined or receiving intervention
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HD036801-Pravastatin; 5U10HD036801-20 (NIH)
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Preeclampsia; Obstetric Labor Complications; Hypertension in Pregnancy
Keywords: Pregnancy; Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia; Obstetric Labor Complications; Hypertension, Pregnancy-Induced | interventions — Pravastatin

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled multi-center clinical trial of 1,550 women with a prior history of preeclampsia that required delivery at less than or equal to 34 weeks 0 days gestation, randomized to one of two arms at participating Maternal Fetal Medicine Units Network clinical centers.
  * 20 mg pravastatin daily
  * Identical appearing daily placebo
Who Masked: Participant, Investigator
Masking Description: Consenting women will be assigned to pravastatin or placebo in a 1:1 ratio according to a randomization sequence prepared and maintained centrally by the Data Coordinating Center (DCC). The two study medication arms of the study (pravastatin or placebo) are double masked; neither the patient nor the clinical staff will be aware of the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pravastatin (Experimental): 20 mg pravastatin daily
  Interventions: Drug: Pravastatin
- Placebo (Placebo Comparator): Identical appearing daily placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pravastatin — 20 mg Pravastatin taken daily
  Arms: Pravastatin
Other: Placebo — Identical appearing placebo pill
  Arms: Placebo

SUMMARY:
This study is a double-blind randomized placebo-controlled trial of 1,550 high-risk women to assess whether daily treatment with pravastatin administered early in pregnancy reduces the rate of a composite outcome of preeclampsia, fetal loss and maternal death. Women with a prior history of preeclampsia with preterm delivery less than 34 weeks will be randomized to pravastatin or placebo daily until delivery. Women will have monthly study visits during pregnancy, a follow-up visit at 6 weeks postpartum and children will have follow-up visits at 2 and 5 years of age.

DETAILED DESCRIPTION:
Preeclampsia complicates approximately 3% to 5% of pregnancies and remains a major cause of maternal and neonatal morbidities and mortality. Women who experience preeclampsia in one pregnancy are at higher risk of developing preeclampsia in a subsequent pregnancy than those who have never experienced the condition. There is evidence from laboratory studies and clinical trials, as well as biological plausibility, to suggest that statins may prevent the development of preeclampsia by reversing various pathways associated with preeclampsia. Pravastatin has a favorable safety profile and pharmacokinetic properties.

The study is a randomized placebo-controlled multi-center clinical trial of 1,550 women with a prior history of preeclampsia that required delivery at less than 34 weeks, randomized to either 20mg pravastatin or an identical appearing placebo daily until delivery. Women with a singleton or twin gestation will be randomized between 12 weeks 0 days and 16 weeks 6 days will be followed monthly during pregnancy and then at 6 weeks postpartum. Children will have follow-up visits at 2 and 5 years of age to assess growth, cognition, behavior, motor skills, vision and hearing.

ELIGIBILITY:
Inclusion Criteria:

1. 16 years or older at time of consent with ability to give informed consent
2. Single or twin gestation with cardiac activity in one or both fetuses. Higher order multifetal gestations reduced to twins, either spontaneously or therapeutically, are not eligible unless the reduction occurred by 13 weeks 6 days project gestational age.
3. Gestational age at randomization between 12 weeks 0 days and 16 weeks 6 days based on clinical information and evaluation of the earliest ultrasound.
4. Documented history (by chart or delivery/operative note review) of prior preeclampsia with delivery less than or equal to 34 weeks 0 days gestation in any previous pregnancy. If in the index pregnancy, the woman was induced by 34 weeks 0 days gestation and delivered within 48 hours in the same hospitalization, that woman would be eligible.
5. Normal serum transaminase (AST/ALT) concentrations documented in the last 6 months.

Exclusion Criteria:

1. Monoamniotic gestation because of the risk of fetal demise
2. Known chromosomal, genetic or major malformations
3. Fetal demise or planned termination of pregnancy. Selective reduction by 13 weeks 6 days gestation, from triplets to twins or twins to singleton is not an exclusion.
4. Contraindications for statin therapy:

   1. Hypersensitivity to pravastatin or any component of the product
   2. Active liver disease: acute hepatitis or chronic active hepatitis
5. Statin use in current pregnancy
6. Patients with any of the following medical conditions:

   1. Uncontrolled hypothyroidism with a TSH level above 10 mIU/L, because of increased risk of myopathy
   2. HIV positive, because of increased risk of myopathy with use of protease inhibitors
   3. Chronic renal disease with baseline serum creatinine ≥1.5 mg/dL, because of association with adverse pregnancy outcomes
7. Current use of concomitant medication with potential for drug interaction with statins (i.e.,, cyclosporine, fibrates, niacin, erythromycin). Patients will not be excluded if the drug is discontinued (at least one week) prior to randomization.
8. Participating in another intervention study that influences the primary outcome in this study
9. Plan to deliver in a non-network site
10. Participation in this trial in a previous pregnancy. Patients who were screened in a previous pregnancy, but not randomized, do not have to be excluded.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2024-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maged Costantine, MD, Principal Investigator — Ohio State University; Monica Longo, MD, PHD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Rebecca Clifton, PhD, Principal Investigator — The George Washington University Biostatistics Center; Victoria Pemberton, RNC, MS, CCRC, Study Director — National Heart, Lung, and Blood Institute (NHLBI)
Locations (12):
- United States (12):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Case Western Reserve-Metro Health, Cleveland, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Given enrollment was limited to 50 participants, the dataset will not be shared.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Costantine MM, Cleary K, Hebert MF, Ahmed MS, Brown LM, Ren Z, Easterling TR, Haas DM, Haneline LS, Caritis SN, Venkataramanan R, West H, D'Alton M, Hankins G; Eunice Kennedy Shriver National Institute of Child Health and Human Development Obstetric-Fetal Pharmacology Research Units Network. Safety and pharmacokinetics of pravastatin used for the prevention of preeclampsia in high-risk pregnant women: a pilot randomized controlled trial. Am J Obstet Gynecol. 2016 Jun;214(6):720.e1-720.e17. doi: 10.1016/j.ajog.2015.12.038. Epub 2015 Dec 23. PMID 26723196

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial began under an FDA clinical hold that limited recruitment to 50 participants of the planned 1,550. The hold was not lifted and the trial was terminated after enrollment of the first 50 participants. We conducted the trial at 13 hospitals. Mothers were enrolled in pregnancy and their offspring followed for 2 years. Recruitment period was Jul 2019 to Dec 2020. Infants were enrolled but were not consented. Two mothers delivered twins resulting in 52 fetus/neonates (26 in each arm).
Groups:
- Pravastatin - Fetus/ Neonates /Infants: Fetus/Neonates/Infants of participants in the 20 mg Pravastatin group
- Placebo - Fetus/ Neonates /Infants: Fetus/Neonates /Infants of participants in the placebo group
Period: Overall Study
Arm/Group | Pravastatin | Placebo | Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Started | 25 | 25 | 26 | 26
Completed | 25 | 25 | 19 | 18 (For the twin gestation in the placebo group, both twins were followed (n=18), however in the analyses, the worst outcome for the twin pair was reported (n=17).)
Not Completed | 0 | 0 | 7 | 8
Not completed — Death | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 4 | 4
Not completed — refused follow-up | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are for the pregnant mothers only as the offspring were not born at the time of randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pravastatin | Placebo | Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants | Total
Number analyzed (Participants) | 25 | 25 | 0 | 0 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline characteristics are for the pregnant mothers only as the offspring were not born at the time of randomization.
  years | 31.6 (4.7) | 31.6 (6.8) |  |  | 31.6 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics are for the pregnant mothers only as the offspring were not born at the time of randomization.
  Participants
    Female | 25 | 25 |  |  | 50
    Male | 0 | 0 |  |  | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline characteristics are for the pregnant mothers only as the offspring were not born at the time of randomization.
  Participants
    American Indian/Alaskan Native | 1 | 0 |  |  | 1
    Asian | 0 | 2 |  |  | 2
    Hispanic | 9 | 8 |  |  | 17
    Native Hawaiian / Pacific Islander | 0 | 0 |  |  | 0
    Non-Hispanic Black | 4 | 6 |  |  | 10
    Non-Hispanic White | 11 | 9 |  |  | 20
    More than 1 self-reported race | 0 | 0 |  |  | 0
Chronic Hypertension [Count of Participants; unit: Participants] — Population: Baseline characteristics are for the pregnant mothers only as the offspring were not born at the time of randomization.
  Participants | 13 | 10 |  |  | 23
Twin pregnancy [Count of Participants; unit: Participants] — Population: Baseline characteristics are for the pregnant mothers only as the offspring were not born at the time of randomization.
  Participants | 1 | 1 |  |  | 2
Gestational age at randomization [Median (Full Range); unit: weeks] — Observed gestational age at randomization Population: Baseline characteristics are for the pregnant mothers only as the offspring were not born at the time of randomization.
  weeks | 14.1 [12.0 to 16.9] | 15.4 [12.0 to 16.9] |  |  | 14.9 [12.0 to 16.9]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Composite of Preeclampsia, Fetal Loss and Maternal Death
Description: Proportion of participants demonstrating a composite of preeclampsia, fetal loss, or maternal death.
  1. Baseline Normotensive: a) Severe hypertension (HTN) or b) Mild HTN w/ any of the following: i.) New-onset proteinuria or doubling in protein w/ baseline proteinuria ii.) Thrombocytopenia iii.) Progressive renal insufficiency iv). Impaired liver function v.) Pulmonary edema vi.) New-onset & persistent cerebral or visual symptoms
  2. Baseline chronic HTN: any of the following a)Severe HTN b) New onset proteinuria or doubling in protein from baseline proteinuria c)Thrombocytopenia d) Progressive renal insufficiency e) Impaired liver function f) Pulmonary edema g) New-onset & persistent cerebral or visual symptoms.
  3. HELLP a) Hemolysis AND b)Thrombocytopenia AND c) AST/ALT ≥ 70 IU/L
  4. Atypical HELLP an occurrence of 2 of the 3: a) Hemolysis, b)Thrombocytopenia, OR c) AST/ALT ≥ 70 IU/L
  5. Eclampsia
  6. Competing outcomes: maternal death before delivery or fetal loss < 20wks, 0 days
Time Frame: 48 hours postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 25 | 25
Participants | 10 | 15
Statistical Analysis 1: Comparison: Pravastatin vs Placebo; Test type: Superiority; Risk Ratio (RR) = 0.67, 95% CI 2-sided [0.37 to 1.19]

2. Secondary Outcome: Proportion of Participants With Preeclampsia With Severe Features
Description: Preeclampsia with severe features as defined by the American College of Obstetricians and Gynecologists (ACOG) diagnostic criteria (i.e., severe hypertension, thrombocytopenia, impaired liver function, progressive renal insufficiency, pulmonary edema, new-onset and persistent cerebral or visual symptoms)
Time Frame: 48 hours postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 25 | 25
Participants | 2 | 4
Statistical Analysis 1: Comparison: Pravastatin vs Placebo; Test type: Superiority; Risk Ratio (RR) = 0.50, 95% CI 2-sided [0.07 to 2.67]

3. Secondary Outcome: Proportion of Participants With Gestational Hypertension
Description: Defined as new onset hypertension in the absence of accompanying proteinuria or other features of preeclampsia
Time Frame: 48 hours postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 25 | 25
Participants | 3 | 1
Statistical Analysis 1: Comparison: Pravastatin vs Placebo; Test type: Superiority; Risk Ratio (RR) = 3.00, 95% CI 2-sided [0.32 to 77.16]

4. Secondary Outcome: Proportion of Participants With Pregnancy Associated Hypertension
Description: Defined as gestational hypertension or preeclampsia
Time Frame: 48 hours postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 25 | 25
Participants | 5 | 9
Statistical Analysis 1: Comparison: Pravastatin vs Placebo; Test type: Superiority; Risk Ratio (RR) = 0.56, 95% CI 2-sided [0.22 to 1.43]

5. Secondary Outcome: Proportion of Participants With Postpartum Preeclampsia
Description: Preeclampsia that occurs more than 48 hours after birth
Time Frame: 48 hours postpartum through 6 weeks post partum
Measure: Count of Participants; unit: Participants
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 25 | 23
Participants | 1 | 0
Statistical Analysis 1: Comparison: Pravastatin vs Placebo; Test type: Superiority; RR not reported given zero events in the placebo group

6. Secondary Outcome: Proportion of Participants With Gestational Diabetes
Description: Gestational diabetes mellitus
Time Frame: At any time during pregnancy through delivery (up to approximately 30 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 25 | 25
Participants | 7 | 4
Statistical Analysis 1: Comparison: Pravastatin vs Placebo; Test type: Superiority; Risk Ratio (RR) = 1.75, 95% CI 2-sided [0.58 to 5.24]

7. Secondary Outcome: Rate of Adherence to Study Medication
Description: Adherence to the medication regimen for the study (daily pill) defined as the time from randomization to delivery. The earliest gestational age at randomization is 12 weeks and most women deliver by 42 weeks gestation which is why the time frame is up to a maximum of approximately 30 weeks. Given the earlier gestational age of delivery in this cohort, the time period is shorter than 30 weeks.
Time Frame: Randomization to delivery (up to approximately 30 weeks)
Measure: Median (Full Range); unit: percentage of compliance
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 25 | 25
percentage of compliance | 88.8 [0 to 100] | 90.3 [0 to 100]
Statistical Analysis 1: Comparison: Pravastatin vs Placebo; Test type: Superiority; p = 0.92, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Proportion of Participants With Severe Maternal Morbidity Composite
Description: A composite of severe maternal morbidity of either maternal death, eclampsia, HELLP syndrome, cerebral vascular accident, heart failure, myocardial infarction, acute respiratory distress syndrome requiring mechanical ventilation, disseminated intravascular coagulopathy, pulmonary edema, renal failure, liver rupture, or placental abruption
Time Frame: Randomization through 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 25 | 25
Participants | 0 | 0
Statistical Analysis 1: Comparison: Pravastatin vs Placebo; Test type: Superiority; RR not reported given zero events in the pravastatin and placebo groups

9. Secondary Outcome: Length of Maternal Hospital Stay
Description: Length of maternal hospital stay for the delivery admission (admission to discharge)
Time Frame: Delivery admission through discharge from the hospital (a median of 3 days)
Measure: Median (Full Range); unit: days
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 25 | 25
days | 3 [1 to 10] | 3 [1 to 44]
Statistical Analysis 1: Comparison: Pravastatin vs Placebo; Test type: Superiority; p = 1.0, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Rate of Adverse Events of Special Interest (AESI) or Serious AESI
Description: Adverse events of Special Interest (AESI) including myalgia and muscle weakness, and serious AESI include maternal myositis, myopathy, rhabdomyolysis, or serious liver injury
Time Frame: Randomization through 48 hours postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 25 | 25
Participants | 1 | 0
Statistical Analysis 1: Comparison: Pravastatin vs Placebo; Test type: Superiority; RR not reported given zero events in the placebo group

11. Secondary Outcome: Gestational Age at Delivery
Description: Gestational age at the time of delivery
Time Frame: Delivery
Population: For twin gestation, the worst outcome for the twin pair is analyzed/reported.
Measure: Median (Full Range); unit: weeks
Groups:
- 20mg Pravastatin - Fetus/ Neonates /Infants: Fetus/Neonates/Infants of participants in the 20 mg Pravastatin group
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 25 | 25
weeks | 36.7 [29.0 to 39.9] | 37.0 [16.3 to 39.4]
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Proportion of Participants With Preterm Birth < 37 Weeks
Description: Preterm birth before 37 weeks gestation
Time Frame: Delivery before 37 weeks
Population: For twin gestation, the worst outcome for the twin pair is analyzed/reported.
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 25 | 25
Participants | 14 | 11
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; Risk Ratio (RR) = 1.27, 95% CI 2-sided [0.73 to 2.23]

13. Secondary Outcome: Proportion of Participants With Indicated Preterm Birth < 37 Weeks
Description: Indicated preterm birth less than 37 weeks
Time Frame: Delivery before 37 weeks
Population: For twin gestation, the worst outcome for the twin pair is analyzed/reported.
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 25 | 25
Participants | 9 | 7
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; Risk Ratio (RR) = 1.29, 95% CI 2-sided [0.57 to 2.91]

14. Secondary Outcome: Proportion of Participants With Preterm Birth < 34 Weeks
Description: Preterm birth before 34 weeks gestation
Time Frame: Delivery before 34 weeks
Population: For twin gestation, the worst outcome for the twin pair is analyzed/reported.
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 25 | 25
Participants | 4 | 7
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; Risk Ratio (RR) = 0.57, 95% CI 2-sided [0.19 to 1.71]

15. Secondary Outcome: Proportion of Fetal or Neonatal Deaths
Description: Death of the fetus or neonate
Time Frame: randomization (mother) through 28 days of life (neonate)
Population: For twin gestation, the worst outcome for the twin pair is analyzed/reported.
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 25 | 25
Participants | 1 | 2
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; Risk Ratio (RR) = 0.50, 95% CI 2-sided [0.02 to 5.35]

16. Secondary Outcome: Birth Weight
Description: Birth weight
Time Frame: Birth
Population: Liveborn neonates only. For twin gestation, the worst outcome for the twin pair is analyzed/reported.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 25 | 23
grams | 2626 (668) | 2543 (884)
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; p = 0.72, t-test, 2 sided

17. Secondary Outcome: Proportion of Small for Gestational Age < 5th Percentile
Description: Birthweight < 5th percentile
Time Frame: Birth
Population: Liveborn neonates only. For twin gestation, the worst outcome for the twin pair is analyzed/reported.
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 25 | 23
Participants | 3 | 2
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; Risk Ratio (RR) = 1.38, 95% CI 2-sided [0.24 to 13.59]

18. Secondary Outcome: Proportion of Small for Gestational Age < 10th Percentile
Description: Birthweight < 10th percentile
Time Frame: Birth
Population: Liveborn neonates only. For twin gestation, the worst outcome for the twin pair is analyzed/reported.
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 25 | 23
Participants | 7 | 6
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.42 to 2.73]

19. Secondary Outcome: Proportion of NICU/Intermediate Nursery Admission
Description: Admission to the neonatal intensive care unit (NICU) or intermediate nursery
Time Frame: Birth through hospital discharge (an average of 4 days)
Population: Liveborn neonates only. For twin gestation, the worst outcome for the twin pair is analyzed/reported. Data missing for 1 pravastatin and 1 placebo participant.
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 24 | 22
Participants | 11 | 9
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; Risk Ratio (RR) = 1.12, 95% CI 2-sided [0.58 to 2.18]

20. Secondary Outcome: NICU/Intermediate Nursery Length of Stay
Description: Length of stay in the neonatal intensive care unit (NICU) and/or intermediate nursery.
Time Frame: Birth through hospital discharge (an average of 4 days)
Population: Neonates admitted to the NICU. For twin gestation, the worst outcome for the twin pair is analyzed/reported.
Measure: Median (Full Range); unit: days
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 11 | 9
days | 13 [2 to 83] | 42 [3 to 220]
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Proportion of Neonates Needing Mechanical Ventilation or Continuous Positive Airway Pressure (CPAP)
Description: Mechanical ventilation or CPAP support
Time Frame: Birth through hospital discharge (an average of 4 days)
Population: Liveborn neonates only. For twin gestation, the worst outcome for the twin pair is analyzed/reported. Data missing for 1 pravastatin and 2 placebo participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 24 | 21
Participants | 7 | 4
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; Risk Ratio (RR) = 1.53, 95% CI 2-sided [0.52 to 4.51]

22. Secondary Outcome: Proportion of Neonates Needing Oxygen Support
Description: Provision of oxygen support for the neonate
Time Frame: Birth through hospital discharge (an average of 4 days)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 24 | 21
Participants | 6 | 4
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; Risk Ratio (RR) = 1.31, 95% CI 2-sided [0.42 to 5.00]

23. Secondary Outcome: Proportion of Neonates With Respiratory Distress Syndrome
Description: Respiratory distress syndrome (RDS), defined as the presence of clinical signs of respiratory distress (tachypnea, retractions, flaring, grunting, or cyanosis), with an oxygen requirement and confirmed by a chest x-ray
Time Frame: Birth through hospital discharge (an average of 4 days)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 24 | 22
Participants | 3 | 4
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; Risk Ratio (RR) = 0.69, 95% CI 2-sided [0.11 to 2.95]

24. Secondary Outcome: Proportion of Neonates With Bronchopulmonary Dysplasia
Description: Bronchopulmonary dysplasia (BPD), defined as oxygen requirement at 28 days of life and at 36 weeks corrected gestational age
Time Frame: 28 days of life and 36 weeks corrected gestational age
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 24 | 22
Participants | 0 | 0
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; RR not reported given zero events in both groups

25. Secondary Outcome: Proportion of Neonates With Necrotizing Enterocolitis
Description: Necrotizing enterocolitis (NEC), defined as modified Bell Stage 2 (clinical signs and symptoms with pneumatosis intestinalis on radiographs) or Stage 3 (advanced clinical signs and symptoms, pneumatosis, impending or proven intestinal perforation)
Time Frame: Birth through hospital discharge (an average of 4 days)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 24 | 22
Participants | 0 | 1
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; RR not reported given zero events in the pravastatin group

26. Secondary Outcome: Proportion of Neonates With Intraventricular Hemorrhage
Description: Intraventricular hemorrhage (IVH) grade III-IV
Time Frame: Birth through hospital discharge (an average of 4 days)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 24 | 22
Participants | 0 | 0
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; RR not reported given zero events in both groups

27. Secondary Outcome: Proportion of Neonates With Periventricular Leukomalacia (PVL)
Description: Periventricular leukomalacia (PVL), diagnosed by neuroimaging
Time Frame: Birth through hospital discharge (an average of 4 days)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 24 | 22
Participants | 0 | 0
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; RR not reported given zero events in both groups

28. Secondary Outcome: Proportion of Neonates Experiencing Early Onset Sepsis
Description: Neonatal sepsis (within first 72 hours after birth). The diagnosis of sepsis will require the presence of a clinically ill infant in whom systemic infection is suspected with a positive blood, cerebral spinal fluid (CSF), or catheterized/suprapubic urine culture; or, in the absence of positive cultures, clinical evidence of cardiovascular collapse or an unequivocal radiograph confirming infection.
Time Frame: Birth to 72 hours from birth
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 24 | 22
Participants | 0 | 0
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; RR not reported given zero events in both groups

29. Secondary Outcome: Proportion of Neonates Experiencing Late Onset Sepsis
Description: Neonatal sepsis (>72 hours after birth). The diagnosis of sepsis will require the presence of a clinically ill infant in whom systemic infection is suspected with a positive blood, cerebral spinal fluid (CSF), or catheterized/suprapubic urine culture; or, in the absence of positive cultures, clinical evidence of cardiovascular collapse or an unequivocal radiograph confirming infection.
Time Frame: Birth through hospital discharge (an average of 4 days)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 24 | 22
Participants | 0 | 1
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; RR not reported given zero events in pravastatin group

30. Secondary Outcome: Proportion of Neonates With Retinopathy of Prematurity
Description: Retinopathy of prematurity (ROP) stage III or higher
Time Frame: Birth through hospital discharge (an average of 4 days)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 24 | 22
Participants | 0 | 0
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; RR not reported given zero events in both groups

31. Secondary Outcome: Proportion of Neonates With Composite Neonatal Outcome
Description: Fetal or neonatal death, RDS, Grade III-IV IVH, PVL, Stage 2 or 3 NEC, BPD, Stage III or higher ROP, or early onset sepsis
Time Frame: Birth through hospital discharge (an average of 4 days)
Population: For twin gestation, the worst outcome for the twin pair is analyzed/reported. Data missing for 1 placebo participant.
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 25 | 24
Participants | 4 | 6
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; Risk Ratio (RR) = 0.64, 95% CI 2-sided [0.17 to 2.04]

32. Secondary Outcome: Proportion of Neonates Experiencing Seizures
Description: Neonatal seizure activity
Time Frame: Birth through hospital discharge (an average of 4 days)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 24 | 22
Participants | 0 | 0
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; RR not reported given zero events in both groups

33. Secondary Outcome: Proportion of Neonates With a Congenital Anomaly / Birth Defect
Description: Congenital anomaly or birth defect excluding any conditions that must have been present before randomization
Time Frame: Randomization through delivery (up to approximately 30 weeks)
Population: For twin gestation, the worst outcome for the twin pair is analyzed/reported. Data missing for 1 placebo participant.
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 25 | 24
Participants | 1 | 1
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.03 to 31.79]

34. Secondary Outcome: Neonatal Auditory Brain Stem Response (ABR)/Otoacoustic Emissions (OAE)
Description: Neonatal auditory brain stem response (ABR)/Otoacoustic Emissions (OAE) test results of fail/refer.
Time Frame: Birth through hospital discharge (an average of 4 days)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 24 | 22
Participants | 0 | 0
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; RR not reported given zero events in both groups

35. Secondary Outcome: BMI for Age at 24 Corrected Months
Description: Body mass index for age percentile at 24 corrected months using Centers for Disease Control (CDC) pediatric growth charts
Time Frame: 24 months of age
Measure: Median (Full Range); unit: percentile
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 16 | 15
percentile | 83.8 [0.3 to 98.7] | 50.6 [0.3 to 96.8]
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney)

36. Secondary Outcome: Cognitive Standard Score From the Bayley Certified Scales of Infant Development III Edition at 24 Months of Age
Description: Bayley Certified Scales of Infant Development III Edition standard score for cognitive abilities at 24 months of age.
  Composite standard scores are derived for cognitive, language, and motor development and scaled to a metric, with a mean of 100, standard deviation of 15, and range of 40 to 160.
  Higher scores mean better outcome.
Time Frame: 24 months of age
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 16 | 14
score on a scale | 93.8 (10.2) | 87.9 (14.6)
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; p = 0.21, t-test, 2 sided

37. Secondary Outcome: Motor Standard Score From the Bayley Certified Scales of Infant Development III Edition at 24 Months of Age
Description: Bayley Certified Scales of Infant Development III Edition standard score for motor abilities at 24 months of age.
  Composite standard scores are derived for cognitive, language, and motor development and scaled to a metric, with a mean of 100, standard deviation of 15, and range of 40 to 160.
  Higher scores mean better outcome.
Time Frame: 24 months of age
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 15 | 13
score on a scale | 90.5 (9.2) | 88.2 (11.9)
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; p = 0.58, t-test, 2 sided

38. Secondary Outcome: Language Standard Score From the Bayley Certified Scales of Infant Development III Edition at 24 Months of Age
Description: Bayley Certified Scales of Infant Development III Edition standard score for language abilities at 24 months of age.
  Composite standard scores are derived for cognitive, language, and motor development and scaled to a metric, with a mean of 100, standard deviation of 15, and range of 40 to 160.
  Higher scores mean better outcome.
Time Frame: 24 months of age
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 15 | 13
score on a scale | 88.9 (16.7) | 87.8 (20.1)
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; p = 0.88, t-test, 2 sided

39. Secondary Outcome: Gross Motor Function Classification System at 24 Months of Age
Description: Level from the Gross Motor Function Classification System at 24 months of age
  Level I (Handles objects easily and successfully) Level II (Handles most objects, but with somewhat reduced quality and/or speed of achievement) Level III (Handles objects with difficulty) Level IV (Handles a limited selection of easily managed objects in simple actions) Level V (Does not handle objects and has severely limited ability to perform even simple actions)
Time Frame: 24 months of age
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 19 | 17
Participants
  Level I | 18 | 16
  Level II | 1 | 1
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; p = 1.0, Fisher Exact

40. Secondary Outcome: Proportion of Children With Hearing Loss at 24 Months of Age
Description: Hearing loss at 24 months of age
Time Frame: 24 months of age
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 19 | 17
Participants | 0 | 2
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; p = 0.22, Fisher Exact; RR not reported given zero events in the pravastatin group

41. Secondary Outcome: Child Behavior Checklist Total Problems T-Score at 24 Months
Description: Total problems T score from the Child Behavior Checklist (CBCL) at 24 months.
  The Child Behavior Checklist (CBCL) is a survey used to detect behavioral and emotional problems in children. The CBCL is filled out by the caregiver. Each of the 100 questions indicates a behavior for which the caregiver scores as Not True (0), Sometimes True (1), or Often True (2). The scores for all the questions are then summed and evaluated against the normative data/T-scores. The raw total scores are converted to norm-referenced T-scores (mean 50, standard deviation of 10). Lower scores represent better outcomes. A T-score of 64 or higher indicates a clinically significant elevation. Lower scores represent better outcomes.
Time Frame: 24 months of age
Measure: Median (Full Range); unit: T-score
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 19 | 16
T-score | 45 [28 to 53] | 44.5 [30 to 84]
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; p = 0.84, Wilcoxon (Mann-Whitney)

42. Secondary Outcome: Proportion of Children With Vision Problems at 24 Months of Age
Description: Vision problems (severe nearsightedness or farsightedness, and eye movement problems) at 24 months of age
Time Frame: 24 months of age
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
Number analyzed (Participants) | 19 | 17
Participants | 0 | 1
Statistical Analysis 1: Comparison: 20mg Pravastatin - Fetus/ Neonates /Infants vs Placebo - Fetus/ Neonates /Infants; Test type: Superiority; p = 0.47, Fisher Exact; RR not reported given zero events in the pravastatin group

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of randomization to delivery (approximately up to 30 weeks) and delivery through 2 years post-delivery (average of 24 months up to a maximum of 42.9 months). Adverse events were collected for maternal participants and their fetuses/neonates.
Description: Other (not include serious) adverse events were not collected for neonates/infants. One maternal participant did not return after randomization and did not complete side effect forms.
Groups:
- 20mg Pravastatin - Mother: 20 mg pravastatin daily
  Pravastatin: 20 mg Pravastatin taken daily
- Placebo - Mother: Identical appearing daily placebo
  Placebo: Identical appearing placebo pill
Arm/Group | 20mg Pravastatin - Mother | Placebo - Mother | 20mg Pravastatin - Fetus/ Neonates /Infants | Placebo - Fetus/ Neonates /Infants
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/25 | 1/26 | 2/26
Serious Adverse Events (participants affected / at risk) | 4/25 | 5/25 | 5/26 | 5/26
Other Adverse Events (participants affected / at risk) | 12/25 | 11/24 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20mg Pravastatin - Mother (N=25) | Placebo - Mother (N=25) | 20mg Pravastatin - Fetus/ Neonates /Infants (N=26) | Placebo - Fetus/ Neonates /Infants (N=26)
Fetal Demise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Termination (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankyloglossia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suspected fetal abnormality (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypospadias (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Poor glycemic control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poor glycemic control and hyperemesis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poor glycemic control and severe hypertension (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeding difficulty (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bowel enterotomy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hypoxic ischemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine rupture (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cervical insufficiency (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension / preeclampsia (Vascular disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Breast Cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Maternal Death (Breast Cancer) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20mg Pravastatin - Mother (N=25) | Placebo - Mother (N=24) | 20mg Pravastatin - Fetus/ Neonates /Infants (N=0) | Placebo - Fetus/ Neonates /Infants (N=0)
Headache (General disorders) | 7 (7) | 5 (5) | NA | NA
Fatigue (General disorders) | 4 (4) | 3 (3) | NA | NA
Dizziness (General disorders) | 2 (2) | 2 (2) | NA | NA
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | NA | NA
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | NA | NA
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | NA | NA
Muscle Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | NA | NA
Anxiety/nervousness (Psychiatric disorders) | 2 (2) | 2 (2) | NA | NA
Influenza-like Symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT03944512/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT03944512/ICF_001.pdf